CLINICAL TRIAL: NCT06094400
Title: Pain and Stress Detection and Relief in People With Dementia Using Portable EEG Headband: A Feasibility Study
Brief Title: Pain and Stress Detection and Relief in People With Dementia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P0045168
Record Dates: First submitted 2023-10-17; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Dementia; Chronic Pain; Perceived Stress
Keywords: dementia; pain; stress
MeSH Terms: conditions — Dementia; Chronic Pain; Pain | interventions — Meditation

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): 10-mintue headband-guided meditation session via Muse Medication App.
  Interventions: Other: Meditation
- Control (Other): 10-minute resting session
  Interventions: Other: Control

INTERVENTIONS:
Other: Meditation — Participants in the intervention group will be furnished with a tablet incorporating a pre-installed Muse Meditation App and a set of headphones. They can choose their preferred immersive soundscape for the meditation session.
  Arms: Intervention
Other: Control — Participants allocated to the control group will similarly wear the portable EEG headband, but they will receive a rest session without any additional intervention
  Arms: Control

SUMMARY:
The objective of this study is to investigate the feasibility and efficacy of using the portable EEG headband and the headband-guided meditation practices for pain and stress relief in people with dementia in Hong Kong. Additionally, it explores the potential use of the headband as a biomarker for pain and stress in this target group.

DETAILED DESCRIPTION:
This project is a Phase II clinical trial to access the feasibility and efficacy of incorporating portable EEG headband-guided meditation for alleviating pain and stress among people with early and moderate dementia in Hong Kong. Sixty dementia people will be recruited. Participants in the intervention group will wear the EEG headband and engage in 10-minute guided meditation sessions, while the control group will wear the EEG headband and undergo a 10-minute resting session. Efficacy will be evaluated using the Wong-Baker Faces Pain Rating Scale, Perceived Stress Scale, and EEG signals associated with pain and stress. Immediate post-assessment focus group interviews will be conducted to explore caregiver's experiences with the use of portable EEG headbands in this study.

ELIGIBILITY:
Inclusion Criteria:

* People with mild to moderate severe dementia;
* Have chronic pain or have experienced stress for at least six months;
* Be able to communicate and express pain;
* Have no prior experience with any type of meditation training;
* Volunteer to participate in the study and provide written informed consent

Exclusion Criteria:

* Person with other acute or terminal illnesses that may not be able to stay in a home living environment frequently;
* With severe visual or hearing problems that would hinder communication;
* With infectious diseases that could be transmitted by using the headband.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-10-17 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Changes on pain level | Pre-intervention, immediately post-intervention
  Pain detection will be measured by the Wong-Baker Faces Pain Rating Scale. The scale show a series of facial expressions, ranging from a happy face at "0", or "no hurt", to a crying face at 10, indicating "hurts like the worst pain imaginable".

SECONDARY OUTCOMES:
Changes on stress level | Pre-intervention, immediately post-intervention
  Stress level will be measured by the Chinese version of the Perceived Stress Scale. It is a 10-item Likert 5-point scale (0=never, 4=very often). Score ranges from 0-40, with higher scores indicating higher level of perceived stress.

IPD SHARING:
Plan to Share IPD: No